CLINICAL TRIAL: NCT02219997
Title: Functional Benefit With ACRYSOF® Natural Chromophore
Brief Title: Functional Vision With ACRYSOF® IQ IOLs Blue Light Filtration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: ILQ830-P001
Record Dates: First submitted 2014-08-18; First posted 2014-08-19 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Cataract
Keywords: Cataract; Intraocular lens (IOL); AcrySof
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACRYSOF IQ IOL (Experimental): ACRYSOF® IQ IOL with or without clear clip-on glasses worn for 3 hours
  Interventions: Device: Clear clip-on glasses; Device: ACRYSOF® IQ IOL
- Clear IOL (Active Comparator): Clear IOL with or without blue light filter clip-on glasses and clear clip-on glasses, worn in a cross-over fashion, as randomized, for 4 hours total
  Interventions: Device: Clear clip-on glasses; Device: Blue light filter clip-on glasses; Device: Clear IOL

INTERVENTIONS:
Device: Clear clip-on glasses — Clip-on glasses with no blue light filtering properties used as a placebo
Device: Blue light filter clip-on glasses — Clip-on glasses with blue light filtering properties similar to ACRYSOF® IOLs
  Arms: Clear IOL
Device: ACRYSOF® IQ IOL — AcrySof IQ Aspheric Natural IOL Model SN60WF with UV and blue light filtering properties, previously implanted
  Arms: ACRYSOF IQ IOL
Device: Clear IOL — Clear IOL, previously implanted
  Arms: Clear IOL

SUMMARY:
The purpose of this study is to compare the reaction time (as measured by braking reaction time in seconds during simulated driving) under glare and no-glare conditions in subjects implanted with ACRYSOF® IQ intraocular lenses (IOLs) to subjects implanted with clear IOLs. This study will enroll subjects previously implanted with IOLs in both eyes for at least 3 months.

DETAILED DESCRIPTION:
Subjects completed 2 visits to the investigational site.

ELIGIBILITY:
Inclusion Criteria:

* Pseudophakes with ACRYSOF® IQ monofocal IOLs or clear (no blue light filter) IOLs in both eyes for at least 3 months.
* Willing and able to understand and sign an informed consent form.
* Corrected visual acuity (CVA) of 20/40 or better.
* Have a valid driver's license.
* Depth perception of at least 100 arc seconds.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Ocular pathology, degeneration, or media opacity.
* Color vision defect.
* Use of ocular or systemic medications that impact macular pigment density or reaction time, including but not limited to, lutein, zeaxanthin, barbiturates, tranquilizers or amphetamines.
* System conditions affecting connective tissue or sensory-motor coordination.
* Other protocol-specified exclusion criteria may apply.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr Clinical Manager, GCRA-Global Med Affairs, Operations, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 6 study centers located in the US.
Pre-assignment Details: Of the 90 enrolled, 22 subjects were exited prior to reaction testing. This reporting group includes all subjects who were reaction tested (68).
Groups:
- AcrySof IQ IOL: ACRYSOF® IQ IOL with clear clip-on glasses worn for 3 hours
- Clear IOL: BLF First, Then Placebo Filter: Clear IOL with blue light filter clip-on glasses worn first and clear clip-on glasses worn second for 4 hours total
- Clear IOL: Placebo Filter First, Then BLF: Clear IOL with clear clip-on glasses worn first and blue light filter clip-on glasses worn second for 4 hours total
Period: First Filter
Arm/Group | AcrySof IQ IOL | Clear IOL: BLF First, Then Placebo Filter | Clear IOL: Placebo Filter First, Then BLF
Started | 33 | 17 | 18
Completed | 33 | 17 | 18
Not Completed | 0 | 0 | 0
Period: Second Filter
Arm/Group | AcrySof IQ IOL | Clear IOL: BLF First, Then Placebo Filter | Clear IOL: Placebo Filter First, Then BLF
Started | 0 | 17 | 18
Completed | 0 | 17 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who were reaction tested.
Groups:
- Clear IOL: Clear IOL with blue light filter clip-on glasses and clear clip-on glasses, worn in a cross-over fashion, as randomized, for 4 hours total
- Total: Total of all reporting groups
Arm/Group | AcrySof IQ IOL | Clear IOL | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (3.2) | 70.3 (2.8) | 70.6 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Braking Reaction Time From No-glare to Glare
Description: Braking reaction time (time to brake, in seconds) was assessed using a driving simulator in no-glare and glare conditions. The subject was presented with a driving scenario during which an obstruction (car pulling over from either side of the road in a random fashion) was presented. Subjects braked in an attempt to avoid colliding with the obstruction, and the braking reaction time was recorded. The experiment was repeated with a glare source present. Both assessments (no-glare and glare) occurred on the same day. Change in braking reaction time was calculated as glare minus no-glare.
Time Frame: Visit 2, up to Day 30
Population: This analysis population includes subjects who were reaction tested with no major protocol violations (per protocol).
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- AcrySof IQ IOL: ACRYSOF® IQ IOL without filters
- Clear IOL: Clear IOL without filters
Arm/Group | AcrySof IQ IOL | Clear IOL
Number analyzed (Participants) | 33 | 33
seconds | 0.07 (0.12) | 0.15 (0.21)

2. Secondary Outcome: Change in Braking Reaction Time From No-glare to Glare (Clear IOLs)
Description: Braking reaction time (time to brake, in seconds) was assessed using a driving simulator in no-glare and glare conditions. The subject was presented with a driving scenario during which an obstruction (car pulling over from either side of the road in a random fashion) was presented. Subjects braked in an attempt to avoid colliding with the obstruction, and the braking reaction time was recorded. The experiment was repeated with a glare source present. Both assessments (no-glare and glare) occurred on the same day. Change in braking reaction time was calculated as glare minus no-glare. This outcome measure was pre-specified for Clear IOL only.
Time Frame: Visit 2, Up to Day 30
Population: This analysis population is a subset of all randomized subjects with no major protocol violations and had non-missing values at the specific time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Placebo Filter: Clear IOLs with placebo colored clip-on filters
- Blue Light Filter: Clear IOL with clip-on glasses with blue light filtering properties
Arm/Group | Placebo Filter | Blue Light Filter
Number analyzed (Participants) | 32 | 32
seconds | 0.17 (0.16) | 0.16 (0.20)

3. Secondary Outcome: Change in Braking Reaction Time From No-glare to Glare (ACRYSOF® IQ IOL + Placebo Filter; Clear IOL + BLF)
Description: as for outcome 1
Time Frame: Visit 2, Up to Day 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- ACRYSOF IQ IOL + Placebo Filter: ACRYSOF® IQ IOL with clear clip-on glasses with no light filtering properties used as a placebo
- Clear IOL + BLF: Clear IOL with clip-on glasses with blue light filtering properties
Arm/Group | ACRYSOF IQ IOL + Placebo Filter | Clear IOL + BLF
Number analyzed (Participants) | 32 | 32
seconds | 0.12 (0.12) | 0.16 (0.20)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of a subject's participation in the study (up to 30 days).
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational product. AEs are reported as pre-treatment and treatment-emergent (initiation of experimental testing).
Groups:
- Pre-treatment: All subjects from time to consent until initiation of experimental testing
- AcrySof IQ IOL: All subjects implanted with ACRYSOF® IQ IOLs from time of initiation of experimental testing
- Clear IOL: All subjects implanted with Clear IOLs from time of initiation of experimental testing
Arm/Group | Pre-treatment | AcrySof IQ IOL | Clear IOL
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 0/90 | 0/33 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.